CLINICAL TRIAL: NCT04019600
Title: Screening of Pulmonary Hypertension in Methamphetamine Abusers (SOPHMA): Rationale and Design of a Multicenter, Cross-sectional Study
Brief Title: Screening of Pulmonary Hypertension in Methamphetamine Abusers
Acronym: SOPHMA
Status: Suspended | Type: Observational
Why Stopped: Recruitment in out-patient clinic has been suspended due to COVID-19 pandemic
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung-Wah David SIU, Clinical Professor, The University of Hong Kong
Other Study IDs: SOPHMA study protocol_v.1
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Methamphetamine Abuse; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Echocardiography — Demographic data and health risk factors will be collected on day of screening, together with the above tests. Right heart catheterization will be separately arranged in patients with a high echocardiographic probability of PAH. For those with a low-intermediate echocardiographic probability, screening will be repeated within 1 year to ensure true negativity of the original scan.
  Other Names: 12-lead electrocardiogram; Serum sampling for brain natriuretic peptide and other biomarkers; 6-minute walking test

SUMMARY:
Methamphetamine is misuse if classified as a "likely" risk factor for pulmonary arterial hypertension (PAH). Nevertheless the actual prevalence of and a screening strategy for PAH in methamphetamine users have not been established. In this study, the prevalence of PAH will be investigated and its independent risk factors among methamphetamine users will be identified.

DETAILED DESCRIPTION:
Methamphetamine is a potent central nervous system stimulant originally prescribed for individuals with neuropsychiatric diseases. Owing to its highly addictive nature, illicit use has emerged as a major public health problem worldwide. It causes methamphetamine use disorders and also affects cardiovascular (CV) system.

PAH is one of those CV complications and is devastating and often life-threatening. In a subsequent retrospective cohort, patients with idiopathic PAH were found to have a much higher prevalence of prior use of methamphetamine and/or its related compounds, compared with patients with chronic thromboembolic pulmonary hypertension or pulmonary hypertension due to a known associated condition. Although current international guidelines recognize methamphetamines as a "likely" cause of drug-induced PAH, almost nothing is known about its prevalence and incidence amongst methamphetamine users.

Besides, since patients with PAH often remain asymptomatic in the early phase, the diagnosis is often made late in the course of the disease, when most small pulmonary arteries have been obliterated, rendering therapy ineffective. Although the prognosis of patients with methamphetamine-associated PAH appears to be much worse than for those with idiopathic PAH, international guidelines and expert consensus have not considered screening for PAH in asymptomatic methamphetamine users.

This study will apply a current guideline-recommended PAH screening algorithm for systemic sclerosis to a large cohort of unselected methamphetamine users in Hong Kong. The study objectives include: 1) to describe the prevalence of PAH among methamphetamine users using a current guidelines-recommended screening algorithm for PAH in systemic sclerosis; 2) to identify independent risk factors for PAH in methamphetamine users; and 3) to develop a prediction model for PAH in methamphetamine users.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years at enrollment
* report of methamphetamine use in the last 2 years
* diagnosed as amphetamine dependent according to the Diagnostic and Statistical Manual of Mental Disorders (the 5th edition) (DSM-V)(13)
* voluntarily agree to participate by providing written informed consent

Exclusion Criteria:

* failed or refused to provide written informed consent

Reference:

13. Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas 2013;25(2):191-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a history of methamphetamine use followed-up in the participating substance abuse clinic will be identified via the computerized database of the clinical management system.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2022-12-22 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of PAH in methamphetamine users | 3 years
  Diagnosis and subtypes, as well as prevalence of PAH in methamphetamine users

SECONDARY OUTCOMES:
Risk factors of PAH in methamphetamine users | 3 years
  Risk factors and a prediction model for PAH in methamphetamine users

CONTACTS AND LOCATIONS:
Overall Officials: Siu-Han JoJo Hai, MBBS, Principal Investigator — Cardiac Division, the University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided